CLINICAL TRIAL: NCT02146768
Title: A Novel Low-dose-contrast Cardiac Computed Tomography Method for Pre-Procedural Guidance in Transcatheter Aortic Valve Replacement
Brief Title: Low-dose-contrast Cardiac Computed Tomography
Acronym: CCTA
Status: Completed | Type: Observational
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 013-234
Record Dates: First submitted 2014-03-03; First posted 2014-05-26 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
Low-dose-contrast CCTA can effectively and safely assess the aortic valve apparatus, and effectively direct the trans-catheter heart valve (THV) size selection by providing accurate annulus sizing, and provide adequate pre-procedural risk-stratification guidance for TAVR/TAVI.

DETAILED DESCRIPTION:
A. INTENT AND PURPOSE

Background:

Optimizing procedural and patient outcomes relies heavily on tomographic imaging data guidance for patients being evaluated for trans-catheter aortic valve replacement or implantation (TAVR) by providing accurate information of the aortic valve apparatus (aortic annulus and its pertinent neighboring structures).

The aortic valve annulus is a dynamic complex elliptical or ovoid 3D entity that is also subject to constant shape deformation across the cardiac cycle in addition to being influenced by the thoracic and intra-thoracic anatomy or variations. Given this inherent nature of the aortic valve annulus, electrocardiographic gated cardiac computed tomographic angiography (CCTA), a robust dynamic 3-dimensional imaging modality, is now widely accepted as the "gold-standard" for evaluating the aortic valve apparatus (AVA). To maximize the information obtained by CT, imaging needs to be performed with intravenous contrast injection.2 CCTA requires administration of iodinated contrast. The volume of iodinated contrast medium is of concern in many patients because candidates for TAVR frequently have impaired renal function.2 Contrast reduction and adherence to protocols for prevention of contrast-induced nephropathy is recommended.2 For access planning via the ilio-femoral route, some groups have reported direct aortic injection with extremely low volumes of contrast.

Reduction of contrast volumes for CCTA of the AVA can be achieved by using lower flow rates than for coronary CT angiography. Although 5 mL/s is typically recommended for coronary imaging, 3 mL/s may sometimes be sufficient for imaging patients in the workup for TAVR.2 Though suggested, these CCTA lower flow rates have not been systematically performed and validated in a population being evaluated for candidacy for TAVR. And as recommended by guidelines, a standard bolus of 80 mL to 120 mL of low-osmolar iodinated contrast is usually necessary for optimal TAVR CCTA scanning.1 In these patients, reducing the dose of iodinated contrast at the time of CCTA acquisition in an attempt to minimize renal injury, and at the same time being able to accurately assess the aortic annulus apparatus (AVA) will be of paramount importance. Some reduction of contrast nephropathy can be accomplished by minimizing contrast volume and the use of iso-osmolar or low-osmolar contrast agents. It has been suggested that the contrast volume threshold can be estimated by using the ratio of contrast volume to creatinine clearance. Nephrotoxicity is more likely when the contrast volume/creatinine clearance ratio exceeds 3.7:1.12 And using this, 3.7 x eGFR (estimated glomerular filtration rate) can be set as the maximal contrast dose for an imaging test or invasive procedure.12 14 CCTA acquisition methods Images were acquired with a Brilliance 64-slice CT scanner (Philips Healthcare, Andover, Massachusetts, USA). As per the recommendations on radiation protection in cardiovascular CT by the Society of Cardiovascular Computed Tomography (SCCT), a tube potential of 100 kV will be considered for patients weighing <90 kg or with a body mass index (BMI) <30; whereas a tube potential of 120 kV will be considered for patients weighing >90 kg and with a BMI >30. It will be adjusted, based on each individual patient's size, to the lowest setting that guarantees acceptable image noise for a suitable signal-to-noise ratio (SNR) to perform analysis.15 The patients' eGFR was first calculated using the MDRD (modification of disease in renal diet) GFR formula. The maximal allowable contrast dose for the CCTA was calculated using 3.7 x [(patient's BSA/1.73) x MDRD-eGFR].14 Next, the dose of contrast chosen for the CCTA was < 50% of the maximal allowable contrast dose. The MDRD formula can underestimate the GFR by about 6.2% in patients with chronic kidney disease and by about 29% in healthy individuals, making this an extremely suitable conservative approach for calculating the contrast dosing, with a tendency only to underdose and never to overdose the contrast. With our extensive experience in doing this, we have decreased the total contrast dose for CCTA of the AVA to 45 ml with satisfactory image quality and SNR for post-processing.

Two separate acquisitions (ECG-synchronized for the aortic root and non-gated for the aorta and peripheral vessels) may be preferable to an ECG-synchronized acquisition of the entire volume to reduce the amount of contrast agent.2 A total contrast dose of 45 ml is essential for ECG-synchronized CCTA that utilizes a 64-multislice CT scanner (MSCT) in order to obtain satisfactory image quality and SNR of the aortic root. Depending on the remaining amount of allowable contrast, a decision was then made to perform a non-gated CT of the aorta and peripheral vessels either with no contrast or a low-dose-contrast protocol that we have in place for selectively enhancing the ilio-femoral arterial regions.

The DICOM data will be post-processed by a workstation capable of advanced image processing, manipulation and optimal multi-planar reformatting.

B. CLINICAL HYPOTHESIS AND OBJECTIVES

Hypothesis:

Low-dose-contrast CCTA can effectively and safely assess the aortic valve apparatus, and effectively direct the trans-catheter heart valve (THV) size selection by providing accurate annulus sizing, and provide adequate pre-procedural risk-stratification guidance for TAVR/TAVI.

Study Design:

The proposed investigation is a retrospective cross-sectional study assessing image quality and safety from a renal standpoint between low-dose-contrast CCTA and traditional-dose-contrast, and effectiveness of low-dose-contrast CCTA in analyzing the complex dynamic 3-pronged aortic annulus geometry pre-procedurally in TAVR to improve procedural and patient outcomes. The study cohort will comprise 150 consecutive patients (75 patients who received low-dose contrast matched by body mass index with 75 patients who received traditional dose contrast) seen at THHBP between January 1, 2011 and June 30, 2013.

Statistical Analysis:

The Bland and Altman plot ratios method comparison will be utilized and the graphs displaying a scatter diagram of the ratios plotted against the averages of the SNR of ascending aorta (SNR-AA) obtained with the two different acquisitions (comparing image quality) will be generated. A generalized propensity score (to adjust for pre-operative clinical and non-clinical factors) approach accounting for the matching will be used to account for possible confounding of the association between low and traditional dose groups and annulus area, annulus perimeter, and maximum and minimum annulus diameter measurements. Moreover, adjusted (by the propensity score) Kappa tests, specificity, and sensitivity will be used to assess agreement between low and traditional dose groups. The outcomes are: CT guided successful TAVR deployment; unsuccessful TAVR deployment (moderate-severe paravalvular leak, rupture, valve embolization, mortality); acute renal failure will be defined as a reduction (pre vs post procedure) in renal function as defined by the RIFLE criteria, occurring will be used to assess differences between the study groups.

Sample Size Considerations:

A study cohort of 50 patients enables the detection of a minimum absolute difference of 3% in the primary outcome incidence (power>80) assuming α=0.05, two-sided test.

B1. Personnel Principal Investigator - Ambarish Gopal Sub-Investigators - Deepika Gopal, Paul Grayburn, William Brinkman, David Brown Research coordinators - Molly Mack, Cecile Mahoney, Christine McKibben, Christina Worley, Jessica Jones Epidemiologist - Giovanni Filardo, PhD, MPH Proposal and Protocol Development-Natalie Settele, PA-C B2. Patients will require the following tests/Lab equipment Patients will have received ECG-gated CTA on a 64 slice CT scanner as standard of care treatment B3. Patient Population The study is a retrospective study of 150 consecutive patients > 18 years of age (75 patients who received low-dose contrast matched by body mass index with 75 patients who received traditional dose contrast) seen at THHBP between January 1, 2011 and June 30, 2013. Patients with MDRD eGFR < 25 will be excluded. The cutoff of 25 was chosen as the maximal allowable dose of contrast for eGFR of 25 would be about 90 ml (3.7 x eGFR of 25), and half of that maximal allowable contrast would be 45 ml (the minimum we require to obtain a CCTA with acceptable SNR for post-processing).

B4. Risks There are no risks to subjects as this is a retrospective trial.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age (75 patients who received low-dose contrast matched by body mass index with 75 patients who received traditional dose contrast) seen at THHBP between January 1, 2011 and June 30, 2013

Exclusion Criteria:

* Patients with MDRD eGFR < 25 will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study is a retrospective study of 150 consecutive patients > 18 years of age (75 patients who received low-dose contrast matched by body mass index with 75 patients who received traditional dose contrast) seen at THHBP between January 1, 2011 and June 30, 2013. Patients with MDRD eGFR < 25 will be excluded. The cutoff of 25 was chosen as the maximal allowable dose of contrast for eGFR of 25 would be about 90 ml (3.7 x eGFR of 25), and half of that maximal allowable contrast would be 45 ml (the minimum we require to obtain a CCTA with acceptable SNR for post-processing).
Sampling Method: Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2014-01; Primary Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Number of patients with acute renal failure. | Baseline (pre and post procedure)
  Compare quality and safety of traditional-dose-contrast CCTA versus low-dose-contrast from a renal standpoint, by using serum creatinine and MDRD - eGFR.

CONTACTS AND LOCATIONS:
Overall Officials: Ambarish Gopal, MD, Principal Investigator — Baylor Research Institute
Locations (2):
- United States (2):
  - Center for Advance Cardiac Care, Plano, Texas
  - The Heart Hospital Baylor Plano, Plano, Texas